CLINICAL TRIAL: NCT05452941
Title: A Phase 4 Study Using a Test-Negative Design to Evaluate the Effectiveness of a 20-valent Pneumococcal Conjugate Vaccine Against Vaccine-type Radiologically-confirmed Community-acquired Pneumonia in Adults >/= 65 Years of Age
Brief Title: A Study to Learn About How 20-Valent Pneumococcal Conjugate Vaccine Works in a Real-world Setting
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7471015; 2023-507293-40-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Non-invasive urine specimens will be collected for pneumococcal detection using BinaxNOW® S. pneumoniae and serotype-specific urinary antigen detection assays.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Cases will be defined as participants hospitalized for RAD+CAP in whom the 7 additional serotypes in 20vPnC beyond 13vPnC plus 15C are identified.
  Interventions: Diagnostic Test: Diagnostic test on urine samples
- Control: All other participants who meet study inclusion criteria but for whom 20vPnC serotypes are not identified from any source and all other RAD+CAP of non-pneumococcal etiologies will serve as test-negative controls.
  Interventions: Diagnostic Test: Diagnostic test on urine samples

INTERVENTIONS:
Diagnostic Test: Diagnostic test on urine samples — Testing by BinaxNOW® S. pneumoniae and serotype-specific urine antigen detection (UAD) assays (UAD-1 and UAD-2).

SUMMARY:
The purpose of this study is to learn about how well the 20-valent pneumococcal conjugate vaccine (20vPnC) works against radiologically-confirmed community-acquired pneumonia (RAD+CAP) due to the 7 new serotypes (types of a bacteria called Streptococcus pneumoniae that cause pneumonia) included in 20vPnC vaccine.

This study is seeking participants who:

* are male or female ≥65 years of age.
* are hospitalized with physician suspicion of community acquired pneumonia (CAP).
* have pneumonia confirmed with imaging like a chest x-ray

Participants will be asked to provide demographic and medical history information, and to provide a urine sample that will be used to test for pneumonia caused by specific strains of a bacteria called Streptococcus pneumoniae. We will compare the proportion of participants who have pneumonia caused by specific strains of the bacteria Streptococcus pneumoniae and were previously vaccinated with 20vPnC with the proportion of participants who have pneumonia caused by something other than vaccine type Streptococcus pneumoniae and have been vaccinated with 20vPnC. Participants will actively take part in the study for about 1-2 days. Information on participant's illness and hospitalization details will be collected through day 30 of their hospitalization through medical chart review.

DETAILED DESCRIPTION:
This is an observational test-negative design study in which all study participants are adults ≥65 years of age hospitalized with RAD+CAP at one of the study sites. The only protocol-specified study procedure is a non-invasive urine specimen collection for pneumococcal detection using BinaxNOW® S. pneumoniae and the serotype-specific urinary antigen detection (UAD) assays. Cases and controls will be differentiated by the presence of vaccine serotypes that are identified by any method, including Quellung reaction of pneumococcal isolates obtained from standard of care (SOC) cultures from blood or high-quality respiratory tract specimens, or serotype specific UAD assays performed on urine specimens. The serotype-specific UAD assays, termed UAD-1 and UAD-2, detect the 13 serotypes in 13vPnC (1, 3, 4, 5, 6A/C, 6B/D, 7F/A, 9V/A, 14, 18C/A/ B/ F, 19A, 19F, 23F) (UAD-1) and 11 additional serotypes (2, 8, 9N, 10A/39, 11A/D/F, 12F, 15B/C, 17F/A, 20A/B, 22F/A, 33F/A) (UAD-2). For the primary objective, cases will be defined as participants hospitalized for RAD+CAP in whom the 7 additional serotypes in 20vPnC beyond 13vPnC plus 15C are identified. All other participants who meet study inclusion criteria but for whom 20vPnC serotypes are not identified from any source and all other RAD+CAP of non-pneumococcal etiologies will serve as test-negative controls.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥65 years of age.
2. Hospitalized participant with physician clinical suspicion of CAP with the presence of ≥2 of the following 10 clinical signs or symptoms:

   * fever (oral temperature >38.0°C/100.4°F or tympanic temperature >38.5°C/101.2°F),
   * hypothermia (<35.5°C/95.9°F measured by a healthcare provider)
   * chills or rigors,
   * pleuritic chest pain,
   * new or worsening cough,
   * sputum production,
   * dyspnea (shortness of breath),
   * tachypnea (respiratory rate >20/min),
   * malaise, or
   * abnormal auscultatory findings suggestive of pneumonia (rales or evidence of pulmonary consolidation including dullness on percussion, bronchial breath sounds, or egophony).
3. Has a radiographic finding that is consistent with pneumonia (e.g., pleural effusion, increased pulmonary density due to infection, the presence of alveolar infiltrates [multi-lobar, lobar, or segmental] containing air bronchograms).
4. Capable of giving signed informed consent

Exclusion Criteria:

1. Any participant who develops signs and symptoms of pneumonia after being hospitalized for ≥48 hours (either at the study site, another transferring hospital, or a combination of these).
2. Received any pneumococcal vaccine ≤30 days prior to enrollment.
3. Unable to provide urine specimen (e.g. anuric).
4. Previous enrollment in the study within the past 30 days.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Males and females ages 65 and older hospitalized for suspected community acquired pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 12500 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2027-06-04 (Estimated); Study Completion 2027-06-04 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of 20vPnC against all (invasive + non-invasive) RAD+CAP due to the 7 additional serotypes in 20vPnC beyond 13vPnC plus 15C | 55 months
  Vaccine effectiveness as calculated as 1 minus the odds ratio for 20vPnC vaccination among cases vs. controls multiplied by 100 adjusted for potentially confounding variables

SECONDARY OUTCOMES:
Effectiveness of 20vPnC against non-invasive RAD+CAP due to the 7 additional serotypes in 20vPnC beyond 13vPnC plus 15C | 55 months
  Vaccine effectiveness calculated as 1 minus the OR for 20vPnC vaccination among cases and controls multiplied by 100 adjusted for potentially confounding variables
Effectiveness of 20vPnC against all RAD+CAP due to any 20vPnC serotype plus 6C and 15C | 55 months
  Vaccine effectiveness calculated as 1 minus the OR for 20vPnC vaccination among cases and controls multiplied by 100 adjusted for potentially confounding variables
Effectiveness of 20vPnC against non-invasive RAD+CAP due to any 20vPnC serotype plus 6C and 15C | 55 months
  Vaccine effectiveness calculated as 1 minus the OR for 20vPnC vaccination among cases and controls multiplied by 100 adjusted for potentially confounding variables
Proportion of participants with RAD+CAP due to the 7 additional serotypes in 20vPnC beyond 13vPnC plus 15C, individually and aggregately | 55 months
  The proportion of participants with RAD+CAP who are positive for any of the 7 additional serotypes contained in 20vPnC beyond 13vPnC plus 15C as detected by UAD-2 or culture
The proportion of all RAD+CAP due to any 20vPnC serotype plus 6C and 15C, individually and aggregately | 55 months
  The proportion of participants with RAD+CAP who are positive for any of the serotypes contained in 20vPnC plus 6C and 15C as detected by UAD-1, UAD-2, or culture
The proportion of all RAD+CAP due to any 13vPnC serotype plus 6C, individually and aggregately | 55 months
  The proportion of participants with RAD+CAP who are positive for any of the serotypes contained in 13vPnC plus 6C as detected by either UAD-1 or culture
Among those positive for a serotype detected by serotype-specific UAD, the proportion of participants with any RAD+CAP due to each UAD serotype individually and aggregately | 55 months
  Among those positive for a serotype detected by serotype-specific UAD, the proportion of participants with RAD+CAP who are positive for any of the UAD serotypes as detected by UAD-1, UAD-2, or culture
The proportion of participants with any RAD+CAP due to S. pneumoniae | 55 months
  The proportion of participants with RAD+CAP who have S. pneumoniae identified by culture, BinaxNOW®, or serotype-specific UADs
Clinical characteristics of disease and hospitalization among those with any RAD+CAP due to all 13vPnC and/or 20vPnC serotypes plus 6C and 15C individually and aggregately | 55 months
  In participants with RAD+CAP, the following metrics overall, and among those positive for any of the serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C, or positive for individual serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C:
  • Proportion with PSI Grade I-V
Clinical characteristics of disease and hospitalization among those with any RAD+CAP due to all 13vPnC and/or 20vPnC serotypes plus 6C and 15C individually and aggregately | 55 months
  In participants with RAD+CAP, the following metrics overall, and among those positive for any of the serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C, or positive for individual serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C:
  • Mean, Median, Min, and Max PSI Grade
Clinical characteristics of disease and hospitalization among those with any RAD+CAP due to all 13vPnC and/or 20vPnC serotypes plus 6C and 15C individually and aggregately | 55 months
  In participants with RAD+CAP, the following metrics overall, and among those positive for any of the serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C, or positive for individual serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C:
  • Proportion in ICU
Clinical characteristics of disease and hospitalization among those with any RAD+CAP due to all 13vPnC and/or 20vPnC serotypes plus 6C and 15C individually and aggregately | 55 months
  In participants with RAD+CAP, the following metrics overall, and among those positive for any of the serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C, or positive for individual serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C:
  • Mean, Median, Min, and Max length (in days) of ICU stay
Clinical characteristics of disease and hospitalization among those with any RAD+CAP due to all 13vPnC and/or 20vPnC serotypes plus 6C and 15C individually and aggregately | 55 months
  In participants with RAD+CAP, the following metrics overall, and among those positive for any of the serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C, or positive for individual serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C:
  • Proportion on ventilator and by type of ventilation used
Clinical characteristics of disease and hospitalization among those with any RAD+CAP due to all 13vPnC and/or 20vPnC serotypes plus 6C and 15C individually and aggregately | 55 months
  In participants with RAD+CAP, the following metrics overall, and among those positive for any of the serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C, or positive for individual serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C:
  • Mean, Median, Min, and Max length (in days) of ventilator use
Clinical characteristics of disease and hospitalization among those with any RAD+CAP due to all 13vPnC and/or 20vPnC serotypes plus 6C and 15C individually and aggregately | 55 months
  In participants with RAD+CAP, the following metrics overall, and among those positive for any of the serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C, or positive for individual serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C:
  • Mean, Median, Min, and Max length (in days) of hospital stay
Clinical characteristics of disease and hospitalization among those with any RAD+CAP due to all 13vPnC and/or 20vPnC serotypes plus 6C and 15C individually and aggregately | 55 months
  In participants with RAD+CAP, the following metrics overall, and among those positive for any of the serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C, or positive for individual serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C:
  • Proportion with respiratory rate ≥30 breaths/min
Clinical characteristics of disease and hospitalization among those with any RAD+CAP due to all 13vPnC and/or 20vPnC serotypes plus 6C and 15C individually and aggregately | 55 months
  In participants with RAD+CAP, the following metrics overall, and among those positive for any of the serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C, or positive for individual serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C:
  • Proportion with PaO2/FiO2 ratio ≤250
Clinical characteristics of disease and hospitalization among those with any RAD+CAP due to all 13vPnC and/or 20vPnC serotypes plus 6C and 15C individually and aggregately | 55 months
  In participants with RAD+CAP, the following metrics overall, and among those positive for any of the serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C, or positive for individual serotypes contained in 13vPnC and/or 20vPnC plus 6C and 15C:
  • Proportion with each discharge disposition

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (91):
- United States (66):
  - Kaiser Permanete Baldwin Park, Baldwin Park, California
  - Kaiser Permanete Downey, Downey, California
  - El Centro Regional Medical Center, El Centro, California
  - Kaiser Permanente Fontana Medical Center, Fontana, California
  - University of California San Francisco - Fresno, Fresno, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente, Los Angeles, California
  - Kaiser Permanente West Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente Vaccine Study Center, Oakland, California
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - Kaiser Permanente Ontario Medical, Ontario, California
  - Southern California Permanente Medical Group (SCPMG), Pasadena, California
  - Kaiser Permanente Riverside Medical Center, Riverside, California
  - Kaiser Permanente Roseville Medical Center, Roseville, California
  - Kaiser Permanente South Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente Zion Medical Center, San Diego, California
  - Kaiser Permanente San Diego Medical Center, San Diego, California
  - Kaiser Permanente San Jose Medical Center, San Jose, California
  - Kaiser Permanente Santa Clara Medical Center, Santa Clara, California
  - Kaiser Permanente South San Francisco Medical Center, South San Francisco, California
  - Kaiser Permanente Walnut Creek Medical Center, Walnut Creek, California
  - Hartford Hospital, Hartford, Connecticut
  - Starling Physicians, Hartford, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory Children's Center - Vaccine Research Clinic (ECC-VRC), Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Norton Clark Hospital, Jeffersonville, Indiana
  - Norton Hospital, Louisville, Kentucky
  - Norton Infectious Diseases Institute, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - University of Louisville School of Medicine, Division of Infectious Diseases, Louisville, Kentucky
  - UofL Health, Jewish Hospital, Louisville, Kentucky
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - UofL Health, Mary & Elizabeth Hospital, Louisville, Kentucky
  - Norton Audubon Hospital, Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - Norton Hospital-Pavilion, Norton Healthcare, Louisville, Kentucky
  - UofL Health, Shelbyville Hospital, Shelbyville, Kentucky
  - UofL Health South Hospital, Shepherdsville, Kentucky
  - Ochsner Medical Center - Kenner, Kenner, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension St. John Hospital, Grosse Pointe Woods, Michigan
  - Henry Ford St. John Hospital, Grosse Pointe Woods, Michigan
  - Beaumont Health Center, Royal Oak, Michigan
  - Beaumont Infectious Diseases Research, Royal Oak, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Henry Ford Wyandotte Hospital, Wyandotte, Michigan
  - UNC Hospitals, Chapel Hill, North Carolina
  - ECU Health Medical Center, Greenville, North Carolina
  - The Brody School of Medicine at East Carolina University, ECU Adult Specialty Care, Greenville, North Carolina
  - UNC Hospitals Hillsborough Campus, Hillsborough, North Carolina
  - Summa Health Clinical Research Center - Specialty, Akron, Ohio
  - Summa Health, Akron, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Kaiser Permanente Sunnyside Medical Center, Clackamas, Oregon
  - Memorial Hermann Hospital, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Carilion Clinic, Roanoke, Virginia
- Israel (9):
  - Emek Medical Center, Afula
  - Samson Assuta Ashdod University Hospital, Ashdod
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Campus, Haifa
  - The Edith Wolfson Medical Center, Holon
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan
  - Infectious Diseases Unit Tel-Aviv Sourasky Medical Center, Tel Aviv
- Spain (16):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitarios De Getafe, Getafe, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - CHUVI- Hospital Alvaro Cunqueiro, Vigo, Pontevedra [pontevedra]
  - Hospital Universitari i Politecnic La Fe, Valencia, València
  - Hospital Universitari Vall D´Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario de Valencia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario Doctor Peset, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471015